CLINICAL TRIAL: NCT02807922
Title: Pharmacological Treatment of Insomnia in Palliative Care: A Randomized, Double-blind, Placebo Controlled, Parallel-group, Multicenter Trial Investigating the Short Time Effect of Zopiclone on Self-reported Sleep Quality in Patients With Advanced Cancer Who Use Opioids and Who Report Insomnia
Brief Title: Pharmacological Treatment of Insomnia in Palliative Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SleepRCT_270215; 2015-005306-11 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Sleep; Insomnia
Keywords: Palliative Care; zopiclone
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zopiclone (Active Comparator): Zopiclone six nights
  Interventions: Drug: Zopiclone
- Placebo (Placebo Comparator): Placebo six nights
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zopiclone
  Arms: Zopiclone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Sleep disturbance is frequent in patients with advanced cancer and decreases the tolerability of other symptoms and impairs quality of life. A detailed description of sleep disturbance and its association with other symptoms, and intervention studies on sleep medications are scarce in patients with advanced cancer. A well-designed randomized controlled trial is needed to determine the short time effectiveness of zopiclone on sleep quality, one of the currently available therapies of insomnia, and further to contribute to the clinical management of insomnia in patients with advanced cancer.

DETAILED DESCRIPTION:
The clinical trial is a randomized, double-blind, placebo controlled, parallel-group, multicenter trial investigating the short time effectiveness of zopiclone on self-reported sleep quality in patients with advanced cancer who use opioids and who report insomnia. Patients with advanced cancer who use opioids and who report insomnia are randomized to either a hypnotic, zopiclone (Arm A) or placebo (Arm B) for six nights. For this study zopiclone Actavis 3.75 mg, 5 mg and 7.5 mg (active comparator) and placebo are defined as Investigational Medicinal Products. The initial dose is zopiclone/placebo 3.75 mg/day. Evaluation of sleep quality is performed in the morning after night 2 and 4 with evaluation of sleep quality by using a numerical rating scale 0-10 with the question "Please circle the number that best describes how you feel now" 0= Best sleep, 10= Worst possible sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified malignant disease
2. Presence of metastatic / disseminated disease
3. Presence of insomnia syndrome defined as:

   1. Self-reported difficulty with initiating sleep (greater than 30 minutes to sleep onset) and/or difficulty maintaining sleep (greater than 30 minutes nocturnal waking time); and
   2. Sleep difficulty at least 3 nights per week; and
   3. Sleep difficulty that causes significant impairment of daytime functioning (The patient will be asked if sleep difficulty result in altered daytime function i.e. feeling tired, lack of energy)
4. Able to comply with all study procedures
5. Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

1. On-going treatment or previous treatment (within last 4 weeks) for more than consecutive 3 days with medications given for insomnia
2. Adverse reactions to zopiclone
3. History of substance abuse
4. Concomitant use of rifampicin and erythromycin
5. Any other contraindication listed on the summary of product characteristics of the investigated medicinal product:

   1. Myasthenia gravis
   2. An established diagnosis of Severe impairment of respiratory function
   3. An established diagnosis of Severe hepatic insufficiency.(Child-Pugh grade B or C)
   4. An established diagnosis of sleep apnea
   5. Known hypersensitivity to the drug or to any component in its formulation: Lactose monohydrate, Calcium hydrogen phosphate, Maize starch, Croscarmellose sodium, Magnesium stearate, Titanium dioxide (E 171), Hypromellose, Iron oxide yellow/Iron oxide red (E 172) and Macrogol
6. Unfit for participation for any reason as judged by the investigator
7. Pregnancy or lactation
8. Women of reproductive age not willing or unable to employ an effective method of contraception (sterilization, using IUD or oral contraception)
9. Scheduled surgery within the next week
10. In the need of change in scheduled opioid dose at baseline (study visit 1)
11. Scheduled intravenous administration of chemotherapy during the study period (from baseline to day 8) or intravenous administration of chemotherapy during the last week
12. Change in corticosteroid dose last week before baseline or planned dose change in corticosteroid dose within 7 days from baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Patient-reported sleep quality | Night six (last study night)
  Primary endpoint is patient-reported sleep quality during the final study night (night six) assessed on a numerical rating scale (NRS) 0-10. 0= Best sleep, 10=Worst possible sleep.

SECONDARY OUTCOMES:
Patient reported total sleep time | Night six (last study night)
Patient reported sleep onset latency | Night six (last study night)
  Sleep onset latency (how long (minutes) it takes to fall asleep

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, Principal Investigator — St. Olavs Hospital
Locations (5):
- Norway (5):
  - Sunniva senter for lindrende behandling, Haraldsplass Diakonale sykehus, Bergen
  - sykehuset Levanger, Levanger
  - Helse Sør-Øst RHF, Sykehuset i Telemark,, Skien
  - St. Olavs Hospital, Trondheim
  - Helse Sør-Øst RHF, Sykehuset i Vestfold,, Tønsberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakobsen G, Engstrom M, Paulsen O, Sjue K, Raj SX, Thronaes M, Hjermstad MJ, Kaasa S, Fayers P, Klepstad P. Zopiclone versus placebo for short-term treatment of insomnia in patients with advanced cancer: study protocol for a double-blind, randomized, placebo-controlled, clinical multicenter trial. Trials. 2018 Dec 27;19(1):707. doi: 10.1186/s13063-018-3088-3. PMID 30591073
- [Derived] Jakobsen G, Sjue K, Paulsen O, Kaasa S, Hjermstad MJ, Klepstad P. Zopiclone versus placebo for short-term treatment of insomnia in patients with advanced cancer-a double-blind, randomized placebo-controlled clinical multicenter phase IV trial. Support Care Cancer. 2022 Dec 19;31(1):60. doi: 10.1007/s00520-022-07537-x. PMID 36534165